CLINICAL TRIAL: NCT03515083
Title: Better Outcomes for Anticoagulation Treatment Through Observation of Atrial Rhythm (BOAT OAR)
Brief Title: Better Outcomes for Anticoagulation Treatment Through Observation of Atrial Rhythm
Acronym: BOAT OAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Collaborators: Bristol-Myers Squibb (Industry); AliveCor (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CV185-584
Record Dates: First submitted 2018-04-21; First posted 2018-05-03 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: apixaban; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomized, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental (Experimental): In the experimental group, each patient will be issued an AliveCor Kardia electrocardiogram monitor that is compatible with their smartphone. Patients will be instructed on the use of the monitor at the initial visit with the study nurse. The patient will submit daily electrocardiogram transmission via on online portal. The study nurse may contact them via text message to remind them to submit their recordings, if they forget.
  The remainder of the treatment of the experimental group will be identical to the control group. At the conclusion of the study, the patient will complete their final atrial fibrillation symptom assessment scale. Their smartphone electrocardiogram monitor will be reviewed to ensure that all of the recordings were retrieved successfully.
  Interventions: Device: Alive Cor Kardia mobile electrocardiogram monitor
- Control (No Intervention): Patients in the control group would receive the standard of care treatment for atrial fibrillation, including cardioversion and ablation as indicated. At monthly visits with the study nurse, a smartphone electrocardiogram monitor will be used to record patient's heart rhythm. No other intervention would be performed during the monthly visit. It is necessary to meet the subject at least once per month to receive the previous month's supply of pills and provide them with the next month's supply of pills. If these subjects were met less frequently, it is possible that the previous month's supply of pills might be lost by the end of the study.
  During the study, if the patient is taken off anticoagulation due to medical contraindication or after an ablation, they will continue to be followed monthly but will not receive apixaban medication.

INTERVENTIONS:
Device: Alive Cor Kardia mobile electrocardiogram monitor — Mobile ECG monitor paired with smart phone application
  Arms: Experimental

SUMMARY:
There is a need to determine actual compliance of direct oral anticoagulants and how to improve this to reduce risk of stroke in patients with atrial fibrillation. Mobile health tools have been implemented world-wide in various patient populations as means of reducing cardiovascular risk and improving disease management. Results of these interventions have been mixed with some interventions demonstrating significant improvement while others demonstrated no difference between the intervention group and the control group. More importantly, these studies indicate that implementation of mobile health tools is feasible in various patient populations and it may just be a matter of finding the correct intervention for a given disease state. The aim of this study is to increase awareness of atrial fibrillation as a means of improving compliance with anticoagulant medication.

DETAILED DESCRIPTION:
The primary hypothesis of this study is that patients with atrial fibrillation will have improved compliance with apixaban therapy if they complete a daily measurement of heart rhythm via a smartphone electrocardiogram monitor, as compared to patients managed in a conventional manner.

Primary Endpoint

1. Primary Endpoint 1: is the percent compliance with apixaban therapy as measured by the amount of apixaban medication that was consumed per month. Compliance is defined as "the extent to which a patient acts in accordance with the prescribed interval and dose of a dosing regimen." Percent compliance will be measured as a continuous variable and strict cutoffs for 'compliant' and 'non-compliant' status will not be imposed.

   Secondary Endpoints
2. Secondary Endpoint 1: is the number of deaths from any cause, stroke, and hospitalization for atrial fibrillation and/or congestive heart failure. Given the low numbers of patients in this study, this will be a composite endpoint of all of these outcomes, since there is insufficient sample size to examine each outcome individually.
3. Secondary Endpoint 2: is the self assessment of atrial fibrillation symptom severity through the use of a standardized scale.

While the secondary endpoints are not directly related to the primary endpoint, there is a possibility that the intervention may lead to changes in health maintenance behavior, which may lead to differences in the secondary endpoints. While this study may not be powered to differentiate between these secondary endpoints, if a trend is noted, this may be hypothesis generating for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Non-valvular atrial fibrillation that is either paroxysmal, persistent or permanent
2. CHA2DS2VASc score of 2 or more
3. Eligible for therapy with apixaban for at least 6 months
4. Possession of a smartphone capable of pairing with the AliveCor Kardia cardiac monitor

Exclusion Criteria:

1. Contraindication to anticoagulation with apixaban for at least 6 months
2. No access to a smartphone capable of pairing with the AliveCor Kardia cardiac monitor
3. Unable to provide informed consent for this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
anticoagulation compliance | 12 months
  percent compliance with apixaban therapy

SECONDARY OUTCOMES:
composite of deaths, strokes, and hospitalizations | 12 months
  number of deaths from any cause, stroke, and hospitalization for atrial fibrillation and/or congestive heart failure
AF symptom severity | 12 months
  self assessment of atrial fibrillation symptom severity through the use of a the Atrial Fibrillation Effect on QualiTy of Life (AFEQT) Questionnaire. Section 1 of the scale gathers details about whether or not the patient is symptomatic and how often they are having symptoms. Section 2 is evaluated as a score from 14-98 indicating the total effect of atrial fibrillation on quality of life. Lower values represent a better outcome. Subscales are not combined.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjaya Gupta, MD, Principal Investigator — Saint Luke's Health System
Locations (1):
- Saint Luke's Health System, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cutler TW, Chuang A, Huynh TD, Witt RG, Branch J, Pon T, White R. A retrospective descriptive analysis of patient adherence to dabigatran at a large academic medical center. J Manag Care Spec Pharm. 2014 Oct;20(10):1028-34. doi: 10.18553/jmcp.2014.20.10.1028. PMID 25278325
- [Background] Zhou M, Chang HY, Segal JB, Alexander GC, Singh S. Adherence to a Novel Oral Anticoagulant Among Patients with Atrial Fibrillation. J Manag Care Spec Pharm. 2015 Nov;21(11):1054-62. doi: 10.18553/jmcp.2015.21.11.1054. PMID 26521117
- [Background] Shore S, Carey EP, Turakhia MP, Jackevicius CA, Cunningham F, Pilote L, Bradley SM, Maddox TM, Grunwald GK, Baron AE, Rumsfeld JS, Varosy PD, Schneider PM, Marzec LN, Ho PM. Adherence to dabigatran therapy and longitudinal patient outcomes: insights from the veterans health administration. Am Heart J. 2014 Jun;167(6):810-7. doi: 10.1016/j.ahj.2014.03.023. Epub 2014 Apr 5. PMID 24890529
- [Background] Schulman S, Shortt B, Robinson M, Eikelboom JW. Adherence to anticoagulant treatment with dabigatran in a real-world setting. J Thromb Haemost. 2013 Jul;11(7):1295-9. doi: 10.1111/jth.12241. PMID 23855420
- [Background] McHorney CA, Crivera C, Laliberte F, Nelson WW, Germain G, Bookhart B, Martin S, Schein J, Lefebvre P, Deitelzweig S. Adherence to non-vitamin-K-antagonist oral anticoagulant medications based on the Pharmacy Quality Alliance measure. Curr Med Res Opin. 2015 Dec;31(12):2167-73. doi: 10.1185/03007995.2015.1096242. Epub 2015 Oct 22. PMID 26393483
- [Background] Cramer JA, Roy A, Burrell A, Fairchild CJ, Fuldeore MJ, Ollendorf DA, Wong PK. Medication compliance and persistence: terminology and definitions. Value Health. 2008 Jan-Feb;11(1):44-7. doi: 10.1111/j.1524-4733.2007.00213.x. PMID 18237359
- [Background] Piette JD, List J, Rana GK, Townsend W, Striplin D, Heisler M. Mobile Health Devices as Tools for Worldwide Cardiovascular Risk Reduction and Disease Management. Circulation. 2015 Nov 24;132(21):2012-27. doi: 10.1161/CIRCULATIONAHA.114.008723. PMID 26596977
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035
- [Derived] Tran AT, Okasha OM, Steinhaus DA, Yousuf OK, Giocondo MJ, Ramza BM, Wimmer AP, Gupta SK. Prospective evaluation of the effect of smartphone electrocardiogram usage on anticoagulant medication compliance. J Interv Card Electrophysiol. 2022 Nov;65(2):453-460. doi: 10.1007/s10840-022-01235-8. Epub 2022 May 5. PMID 35513562
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555